CLINICAL TRIAL: NCT05514600
Title: The Impact of Fascial Defect Closure for Minimally Invasive Parastomal Hernia Repair
Brief Title: Fascial Defect Closure for Minimally Invasive Parastomal Hernia Repair
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slower than expected enrollment and early hernia recurrence
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Clayton Petro, MD, FACS, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-634
Record Dates: First submitted 2022-08-06; First posted 2022-08-24 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Parastomal Hernia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascial closure (Active Comparator): This arm will have the parastomal fascial defect closed with a running barbed suture prior to mesh placement.
  Interventions: Procedure: closure of parastomal hernia fascial defect
- No fascial closure (No Intervention): This arm will undergo mesh placement +/- fixation without the fascial defect being closed prior.

INTERVENTIONS:
Procedure: closure of parastomal hernia fascial defect — For subjects randomized to the fascial closure arm, the parastomal defect will be closed using barbed, running suture prior to placement of the mesh.
  Arms: Fascial closure

SUMMARY:
Fascial closure was not originally a routine component of minimally invasive parastomal hernia repairs, but several recent advancements have made fascial closure more common in this context. These include barbed self-locking sutures that aid intracorporeal fascial closure under tension, and wristed instrumentation offered by the robotic platform when available. The investigator aims to characterize the clinical significance of closing the fascia adjacent to the stoma during a MIS parastomal hernia repair.

The investigator hypothesizes that fascial closure will not have a significant impact on postoperative stoma specific quality of life but will reduce long-term recurrence.

DETAILED DESCRIPTION:
This trial will follow the same methodology of data collection employed in previous randomized controlled trials (RCTs) performed by the Cleveland Clinic Center for Abdominal Core Health. The Abdominal Core Health Quality Collaborative (ACHQC) registry will serve as the main platform for data collection. This will be a single-institution study, performed at the Cleveland Clinic Foundation (CCF) hospital in Ohio. Enrollment and surgeries are anticipated to occur at Cleveland Clinic Center for Abdominal Core Health located at Main Campus.

After minimally invasive access and completion of adhesiolysis the surgeon will determine if a minimally invasive intraperitoneal Sugarbaker repair can be achieved. Those patients who cannot be repaired by a minimally invasive intraperitoneal Sugarbaker technique or who convert to an open procedure will be considered screen failures. For those able to be repaired with a minimally invasive intraperitoneal Sugarbaker technique, patients will be randomized to parastomal fascial closure with a running #1 Stratafix symmetric or not. Management of concomitant non-stoma defects that will also be covered with intraperitoneal mesh will be managed at the surgeon's discretion. Surgeons should achieve at least 4cm of mesh overlap from the edge of the parastomal fascial edge before closure. The edge of the mesh can be secured with sutures or tacks at the surgeon's discretion and details will be collected per standard of care in the ACHQC.

Baseline patient demographic information, medical co-morbidities, hernia characteristics, operative details, and 30-day outcomes are already captured within the ACHQC database, allowing for follow-up, and data capture with decreased effort outside of routine care. Baseline patient eligibility criteria will be obtained at initial patient recruitment, and baseline ACHQC questionnaires will be completed following patient consent. Standard of care questionnaires include information on baseline opioid consumption, the PROMIS Pain Intensity instrument, and Hernia Related Quality-of-Life Survey (HerQles). Patients will be required to complete these forms at each clinic visit, or via telephone contact, as this is standard procedure for all patients in our hernia practice. Follow-up will be targeted at 30 +/- 15 days, 1 year ± 4 months, and 2 years ± 6 months with CT scans of the abdomen and pelvis done at the 1 and 2 year time points which is the standard of care for Cleveland Clinic.

Non-standard of care outcome measures, operative time, parastomal defect dimensions (can be separate and distinct in the presence of a concomitant ventral hernia) and randomization will be stored in RedCAP®. Additional tools include the Colostomy Impact Score, which assesses stoma-specific quality of life and will be attained at baseline, 30-days, 1 year, and 2 years. Finally, decision regret using the decision regret scale will be assessed at 30-days, 1 year, and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* End or loop-end stoma with a parastomal defect - candidate for minimally invasive Sugarbaker repair at the discretion of the staff surgeon.
* Anticipated parastomal fascial defect should not exceed 7cm in any direction
* Patient able to tolerate a minimally invasive repair, the surgeon can achieve minimally invasive access and complete a minimally invasive adhesiolysis.
* Bowel able to be lateralized at least 4cm beyond the edge of the parastomal fascial defect

Exclusion Criteria:

* Loop stoma
* Parastomal fascial defect >7cm
* Concomitant ventral defect or complexity of the repair warrants open repair at the discretion of the staff surgeon
* Minimally invasive Sugarbaker repair with intraperitoneal mesh cannot be achieved.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Stoma specific quality of life score (1 year) | 1 year
  The investigators will compare stoma-specific quality of life score using the Colostomy Impact Score (a patient reported survey with 7 questions with a range of 0-38 and higher scores indicating more negative impact on quality of life) at 1 year +/-4 months after minimally invasive Sugarbaker parastomal repair with and without parastomal fascial closure.

SECONDARY OUTCOMES:
Stoma specific quality of life score (30 days) | 30 days
  The investigators will compare stoma-specific quality of life using the Colostomy Impact Score at 30+/-15 days after surgery in both groups. Colostomy Impact score is a patient reported survey with 7 questions with a range of 0-38 and higher scores indicating more negative impact on quality of life.
Stoma specific quality of life score (2 years) | 2 years
  The investigators will compare stoma-specific quality of life using the Colostomy Impact Score at 2 years +/-6 months after surgery in both groups. Colostomy Impact score is a patient reported survey with 7 questions with a range of 0-38 and higher scores indicating more negative impact on quality of life.
Recurrence | 2 years
  The investigators will compare composite parastomal hernia recurrence at 1 year +/- 4 months and 2 years +/- 6 months including patient reported bulge, clinical examination, and CT scan.
Pain Intensity | 2 years
  The investigators will compare Patient Reported Outcomes Measurement Information System (PROMIS Pain Intensity) 3a scores at baseline, 30+/-15 days, 1 year +/- 4 months, and 2 years +/- 6 months. PROMIS is a scale from 30.7- 71.8 with higher numbers indicating higher pain.
Abdominal Wall Specific Quality of Life | 2 years
  The investigators will compare Hernia Related Quality of Life Survey (HerQLes) score at baseline, 30+/-15 days, 1 year +/- 4 months and 2 years +/- 6 months. HerQLes is a 12 question survey with a score that is converted to a numeric score between 0-100, where a higher score indicates better quality of life.
Length of stay | 30 days
  The investigators will compare length of stay in days during the index admission between the two groups.
Ileus | 30 days
  The investigators will compare incidence of ileus, defined as nasogastric tube placement, between the two groups within the first 30+/-15 days after surgery.
Opioid consumption | 30 days
  The investigators will compare opioid consumption in morphine milligram equivalents between the two groups at 30+/-15 days after surgery.
Wound morbidity | 30 days
  The investigators will compare incidence of wound morbidity (including surgical site infection, surgical site occurrence, surgical site occurrence requiring procedural intervention, and reoperation) between the two groups at 30+/-15 days.
Decision Regret | 2 years
  The investigators will compare patient decision regret between the two groups using the Decision Regret Scale (a five question patient reported survey that is scored from 0-100, with lower scores indicate less regret) at 30+/-15 days, 1 year +/-4 months, and 2 years +/- 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided